CLINICAL TRIAL: NCT05363579
Title: A Randomized Controlled Trial (RCT) on the Effectiveness of Tuina in Managing Chronic Low Back Pain
Brief Title: A Study on the Effectiveness of Tuina in Managing Chronic Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Singapore General Hospital (Other)
Collaborators: The Head Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2020/2798
Record Dates: First submitted 2022-03-17; First posted 2022-05-06 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Chronic Low-back Pain
MeSH Terms: interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: This is a randomized, single-blind, parallel-controlled study. The test group is TUINA group and the TUINA combined with PT group, the control group is PT group.
Who Masked: Outcomes Assessor
Masking Description: Only the Principal Investigator would not be blinded. The randomizing scheme will be produced by using statistical analysis software SAS 9.3 with "proc plan" program or excel randomization program to generate the randomization codes. After production, it will be signed and sealed by the Principal Investigator. It will not be allowed to be checked by anyone except the Principal Investigator. Blinded research assessors in each center will be responsible for getting random envelopes from the PI.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Physiotherapy (Other): It is a form of therapy.
  Interventions: Other: Physiotherapy
- Tuina Therapy (Other): It is a form of therapy.
  Interventions: Other: Tuina therapy
- Physiotherapy mixed with Tuina (Other): It is a form of therapy.
  Interventions: Other: Physio and Tuina therapy

INTERVENTIONS:
Other: Physiotherapy — Physiotherapy can be defined as a treatment method that focuses on the science of movement and helps people to restore, maintain and maximize their physical strength, function, motion and overall well-being by addressing the underlying physical issues.
  Arms: Physiotherapy
Other: Tuina therapy — Tuina is mainly applied to the meridians or acupoints by manipulation techniques such as pushing, grasping, pressing and rubbing of the soft tissues or muscles of the body. It is reported to improve circulation and the qi in the body.
  Arms: Tuina Therapy
Other: Physio and Tuina therapy — Physiotherapy mixed with Tuina
  Arms: Physiotherapy mixed with Tuina

SUMMARY:
Low back pain (LBP) is a common clinical symptom prompting patients to seek medical care. 80% of adults experience LBP during their lifetime. The causes of CNLBP are still not fully elucidated and there is currently no gold standard treatment for CNLBP. The mainstay of conservative treatment for CNLBP includes pharmacological interventions, weight loss and physiotherapy.

More recently, Tuina, a component of Traditional Chinese Medicine, has been used to treat CNLBP as well. Tuina is mainly applied to the meridians or acupoints by manipulation techniques such as pushing, grasping, pressing and rubbing of the soft tissues or muscles of the body. It is reported to improve circulation and the qi in the body. However, recent systematic reviews on the efficacy of Tuina in the management of CNLBP were not able to definitively conclude the effectiveness of Tuina due to the poor methodological quality of the studies.

Therefore, this study is a single blind, randomized controlled trial (RCT), which aims to determine the efficacy and safety of Tuina in the management of CNLBP. Similar studies are also conducted in China (First Affiliated Hospital of Jinan University) and USA (Mayo Clinic).

Patients from SGH Orthopaedic clinics with CNLBP, will be recruited for this RCT, and will be randomly divided into 3 intervention groups: Physiotherapy intervention group as the control group, Tuina intervention group, and combined intervention (Tuina + Physiotherapy) group. The intervention will last for 2 months, and follow up assessments will be conducted at the 5th month. Outcome measures include Visual Analog Scale (VAS), Spinal range of motion, Oswestry Disability Index (ODI), TCM Syndrome scale and quality of life 36 item short form survey, (SF-36).

DETAILED DESCRIPTION:
This is a randomised controlled study, single blind with the assessor blinded to the intervention groups of the study.

204 patients (68 per group) with CNLBP will be recruited from the Outpatient Spine Clinic of the Department of Orthopaedic Surgery, SGH, as referred by the Orthopaedic Surgeons.

They will be screened by the assessor, using the inclusion and exclusion criteria listed in K1 and K2 and if consent is given, baseline assessment of the outcomes variables will be conducted. After assessment, the subjects will be randomized into Tuina (TN) group and control physiotherapy (PT) group and Tuina combined physiotherapy (TP) group in a 1:1:1 ratio by the PI. Stratified blocked randomization method will be used in this study. The assessor remainds blind to the treatment groups for all outcome assessments. Standard Physiotherapy and Tuina procedures will be used in the treatment of the subjects according to their presenting symptoms. Education and home exercises will also be taught as appropriate. All subjects will be provided with a maximum of 6 treatment sessions, after which a post-intervention assessment will be conducted.

The intervention that is not standard is the combination of Tuina and Physiotherapy sessions, which is the intervention in Group TP.

Due to the particularity of Tuina and the PT intervention, the operators or intervention providers and the patients are not blinded to the treatment group. The Research Accessors perform the baseline evaluations and follow-up observation, and statistical analysis, hence they will be blinded in this study.

Each group will perform 6 sessions of Interventions over a period of 2 months. However, if the subject improves completely before the completion of the 6 sessions, they need not continue with the remaining sessions.

Criteria for discharge or to discontinue physiotherapy when the subject has improved completely based on the following:

1. Patient able to reach SMART goals set at initial physiotherapy/Tuina visit.
2. Patient feels that he/she is able to manage condition independently.
3. Patient's pain levels are well controlled and/or functional goals have been met.

In all cases, a follow up of the outcome measures will be conducted at the 5th month from the baseline measurement by the blinded assessor.

All interventions will be conducted at the Physiotherapy Department at SGH or at the respective TCM clinics. Physiotherapy procedures conducted are part of the standard care for patients with CNLBP, the Tuina procedures that will be conducted for patients with CNLBP are also part of the standard procedures that are being practiced at the TCM clinic.

MOH Registered TCM practitioners will be recruited by SGH to conduct standard Tuina intervention for this study. A room at the Rehabilitation Centre, SGH, will be provided for the Tuina Practitioners to perform Tuina intervention for the subjects or at the respective TCM clinics at the following locations:

1. Zhongjing TCM Clinic, 36 Hamilton Road, Singapore 209206
2. Aequilibrium TCM, 9 King Albert Park, #02-13, KAP Mall, Singapore 598332

The Physiotherapy intervention is provided by Physiotherapists from the Physiotherapy Department, SGH. All interventions for TCM and PT are provided free for all participants and costs borne by the grant provider.

The criteria for selecting service providers for both TCM and Physiotherapy Practitioners are :

1. Must be registered practictioners with MOH.
2. Have at least one year experience treating patients with low back pain conditions.

The outcome measurements consist of

1. VAS - recording the number from the scale from 0 to 10.
2. Spinal flexion and side/lateral flexion range of motion.
3. Oswestry Disability Index
4. 36- item Short Form Survey or SF 36
5. Traditional Chinese Medicine Syndrome Scale

These measurements will be conducted at the baseline, post intervention at 2 months and follow up at 5 months from baseline by the Research Assessor, who is also a study team member but blind to the intervention group. The Assessor will be trained to conduct the measurements for all subjects, by the study team Physiotherapist and TCM practitioner.

Besides these measurements, other data such as patient demographics, social and medical history and other related treatment session reports, such as duration, frequency, satisfaction and adverse events will also be recorded for analysis where appropriate.

ELIGIBILITY:
Inclusion Criteria:

Voluntary participants aged 21 to 75 years old, regardless of gender, who has CNLBP according to the specific diagnostic criteria below:

1. Pain and discomfort of unknown etiology in the low back region, (with or without referred pain to the lower limbs), lasting for more than 12 weeks.
2. There may be muscle weakness, stiffness, limited mobility or reduced spinal coordination during spinal movement.
3. Physical examination showed an increase in muscle tension or a significant localized tenderness point (trigger point) in the painful area, with negative straight-leg raising test, and no signs of nerve root lesion

Exclusion Criteria:

1. Patients with severe skin diseases (e.g., skin cancer, erysipelas, severe eczema, severe dermatitis, severe psoriasis and severe hives lupus).
2. Recent (within the last month) episodes of spinal pathologies such as fractures, tumors, inflammatory and infectious diseases.
3. History of spine surgery.
4. Recent (within the last month) episodes of cardiovascular or metabolic disorders.
5. Patients diagnosed with psychosocial factors affecting the cognitive and mental faculties such as major depression, moderate to severe dementia and severe psychiatric diseases (such as schizophrenia, bipolar affective disorder, and paranoid psychosis).
6. Women who are Pregnant.
7. Full-time National Service men or on workmen compensation.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Visual Analog Scale at 2 months | From date of randomization until date of first documented progression, up to 60 days
  Recording pain according to number on the scale. Min value is 0 and max value is 10. Higher scores mean worse outcome.
Change from post recruitment 2 months Visual Analog Scale at 5 months | From date of randomization until date of second documented progression, up to 150 days
  Recording pain according to number on the scale. Min value is 0 and max value is 10. Higher scores mean worse outcome.
Change from baseline spinal Range of Motion at 2 months | From date of randomization until date of first documented progression, up to 60 days
  Degree of Spinal flexion and side/lateral flexion range of motion using goniometer and inclinometer
Change from post recruitment 2 months spinal Range of Motion at 5 months | From date of randomization until date of second documented progression, up to 150 days
  Degree of Spinal flexion and side/lateral flexion range of motion using goniometer and inclinometer
Change from baseline Oswestry Disability Index at 2 months | From date of randomization until date of first documented progression, up to 60 days
  A score of 0-20 reflects minimal disability, 21-40 moderate disability, 41-60 severe disability, 61-80 crippled, and 81-100 bed-bound. Higher scores mean worse outcome.
Change from post recruitment 2 months Oswestry Disability Index at 5 months | From date of randomization until date of second documented progression, up to 150 days
  A score of 0-20 reflects minimal disability, 21-40 moderate disability, 41-60 severe disability, 61-80 crippled, and 81-100 bed-bound. Higher scores mean worse outcome.
Change from baseline 36- item Short Form Survey at 2 months | From date of randomization until date of first documented progression, up to 60 days
  The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability.
Change from post recruitment 2 months 36- item Short Form Survey at 5 months | From date of randomization until date of second documented progression, up to 150 days
  The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability.
Change from baseline Traditional Chinese Medicine Syndrome scale at 2 months | From date of randomization until date of first documented progression, up to 60 days
  The presence of a TCM syndrome is diagnosed when the individual syndrome's score is >7. The severity level of the syndrome is further divided into mild (score, 7-14), moderate (score, 15-22), and severe (score ≥23), with 30 being the highest score.
Change from post recruitment 2 months Traditional Chinese Medicine Syndrome scale at 5 months | From date of randomization until date of second documented progression, up to 150 days
  The presence of a TCM syndrome is diagnosed when the individual syndrome's score is >7. The severity level of the syndrome is further divided into mild (score, 7-14), moderate (score, 15-22), and severe (score ≥23), with 30 being the highest score.
Physiotherapy / Tuina treatment satisfaction survey at 2mths | From date of randomization until date of first documented progression, up to 60 days
  Recording satisfaction according to number on the scale. Min value is 0 and max value is 4.

CONTACTS AND LOCATIONS:
Locations (1):
- Singapore General Hospital, Singapore, Singapore